CLINICAL TRIAL: NCT06192953
Title: Early Functional Proprioceptive Stimulation Post-stroke
Acronym: StimProF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-AOI-14
Record Dates: First submitted 2023-12-11; First posted 2024-01-05 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Stroke (CVA) or TIA
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulated group (Experimental): 5 sessions per week for 6 weeks maximum of reeducation with Functional Proprioceptive Stimulation
  Interventions: Other: Functional Proprioceptive Stimulation
- Simulated group (No Intervention): 5 sessions per week for 6 weeks maximum with the device of Functional Proprioceptive Stimulation settled but not activated

INTERVENTIONS:
Other: Functional Proprioceptive Stimulation — Orthoses with a system of 12 stimulators producing mechanical oscillations are attached to the joints of the upper limbs (wrist, elbow and shoulder) or lower limb joints (ankle, knee, hip). These stimulators, which are all synchronized, deliver mechanical oscillations (FPS) that give the illusion of complex movements, while the patient is bedridden, neither moving nor producing effort.
  Arms: Stimulated group

SUMMARY:
The main objective of our study is to evaluate the impact of the use of Functional Proprioceptive Stimulation (FPS) on the recovery of the postural and motor functional capacities of the patient in the subacute phase of a stroke.

The hypothesis is that the use of FPS has a positive impact on the recovery of the patient's functional abilities, as well as on the duration of treatment until the sit/stand transfers are completed.

To evaluate this potential effect,there will be a randomization with two groups : one will have 5 sessions a week for 6 weeks maximum of SPF and the other groupe will have the same sessions but with the device stettled but not activated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient hospitalized at Cimiez University Hospital;
* Ischemic or hemorrhagic cerebrovascular accident (CVA) of less than two weeks;
* Hemiparesis requiring rehabilitation treatment;
* Patient with a SFPASS score ≤ 6;
* Patient affiliated to or beneficiary of a social security scheme;
* Signature of informed consent

Exclusion criteria :

* NIHSS > 20;
* Muscle spasticity of the lower limbs requiring botulinum toxin injection
* Inability to understand rehabilitation instructions;
* Vulnerable people
* Pregnant women, parturients and breastfeeding mothers, persons deprived of their liberty by a judicial or administrative decision, persons hospitalized without consent and persons admitted to a health or social establishment for purposes other than research,
* Adults who are subject to a legal protection measure or who are unable to express their consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Score at the Short Form of Postural Assessment Scale for Stroke Patients (SFPASS) | Inclusion
  The SFPASS is a short instrument used to assess balance in lying, sitting and standing positions. It was designed specifically for stroke patients and is appropriate for all individuals, regardless of their postural performance. SFPASS focuses on mobility in bed and sitting to standing transfer. It is composed of 5 items rated on a 3-point scale with total scores ranging from 0 to 15 and is evaluated by a health professional.
Score at the Short Form of Postural Assessment Scale for Stroke Patients (SFPASS) | Every week during 5 weeks maximum
  The SFPASS is a short instrument used to assess balance in lying, sitting and standing positions. It was designed specifically for stroke patients and is appropriate for all individuals, regardless of their postural performance. SFPASS focuses on mobility in bed and sitting to standing transfer. It is composed of 5 items rated on a 3-point scale with total scores ranging from 0 to 15 and is evaluated by a health professional.
Score at the Short Form of Postural Assessment Scale for Stroke Patients (SFPASS) | 6 weeks
  The SFPASS is a short instrument used to assess balance in lying, sitting and standing positions. It was designed specifically for stroke patients and is appropriate for all individuals, regardless of their postural performance. SFPASS focuses on mobility in bed and sitting to standing transfer. It is composed of 5 items rated on a 3-point scale with total scores ranging from 0 to 15 and is evaluated by a health professional.
Score at the Short Form of Postural Assessment Scale for Stroke Patients (SFPASS) | 10 weeks
  The SFPASS is a short instrument used to assess balance in lying, sitting and standing positions. It was designed specifically for stroke patients and is appropriate for all individuals, regardless of their postural performance. SFPASS focuses on mobility in bed and sitting to standing transfer. It is composed of 5 items rated on a 3-point scale with total scores ranging from 0 to 15 and is evaluated by a health professional.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No